CLINICAL TRIAL: NCT02251379
Title: Environmental Control as Add-on Therapy in Childhood Asthma
Acronym: ECATCh
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NA_00093323
Record Dates: First submitted 2014-09-22; First posted 2014-09-29 (Estimated); Results first posted 2019-11-04 (Actual); Last update posted 2019-11-20 (Actual); Status verified 2019-11

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma | interventions — Fluticasone; Fluticasone-Salmeterol Drug Combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ECS + Medication Group (Experimental): The Environmental Control Strategy ("Home Environmental Intervention") plus inhaled corticosteroids or inhaled corticosteroids plus long-acting beta agonist. (Flovent Diskus or Advair diskus)
  Interventions: Drug: Flovent Diskus; Other: Home Environmental Intervention; Drug: Advair Diskus
- Medication Group Alone (Active Comparator): inhaled corticosteroids or inhaled corticosteroids plus long-acting beta agonist. (Flovent Diskus or Advair diskus)
  Interventions: Drug: Flovent Diskus; Drug: Advair Diskus

INTERVENTIONS:
Drug: Flovent Diskus — Inhaled corticosteroids
  Other Names: Flovent Diskus, 50 mcg, 100mcg, 250 mcg
Other: Home Environmental Intervention — Mouse, Cockroach, Furry pets, Dust mites, Smoking, air purifiers, laundered bedding
  Arms: ECS + Medication Group
Drug: Advair Diskus — inhaled corticosteroids + long-acting beta agonist

SUMMARY:
This study evaluates the effects of adding on an environmental home intervention to standard asthma medication management on controller medication requirements among children and adolescents with asthma. The investigators hypothesize that the addition of an individually-tailored, multi-faceted Environmental Control Strategy (ECS) to guidelines-based controller medication will result in less controller medication requirement and allergic inflammation than controller medication alone among urban asthmatic children.

DETAILED DESCRIPTION:
The study is a parallel arm study of an individually tailored, multi-faceted ECS plus controller medication titration versus controller medication titration alone. After a 4-week run-in period to stabilize the asthma, the investigators will randomize 200 Baltimore children with persistent asthma and a recent exacerbation in a 1:1 ratio to the two arms and follow the children for six months. There will be five clinic visits and three home visits over this time period for clinical and home assessments, respectively. There will be up to four environmental intervention visits for participants randomized to the environmental control plus controller medication group. The environmental modules include mouse, cockroach, furry pets, dust mites, and smoking. Air purifiers and laundered bedding are also included in this arm. Participants randomized to the controller medication group have the option of having one home visit after completing the study at which the participants will receive home intervention services that the environmental control plus controller medication group received. Participants will have repeated assessment of: controller medication requirements; secondary clinical, physiologic, and inflammatory outcomes; and particulate matter (PM), air nicotine, and allergen levels.

ELIGIBILITY:
Inclusion Criteria:

* Have physician-diagnosed asthma at least 1 year prior to the baseline visit, or asthma symptoms for at least 1 year
* Meet criteria for current persistent asthma defined as either:

  1. On a long-term controller medication for asthma, or
  2. Meet National Asthma Education and Prevention Program (NAEPP) guideline requirements for persistent disease:(46)
* Asthma symptoms 3 or more days per week over the past 2 weeks or
* Nocturnal asthma symptoms at least 3 times in the past month
* Have evidence of uncontrolled disease as defined by at least one of the following:

  1. One asthma-related unscheduled visit to an emergency department (ED), clinic or urgent care facility in the previous 12 mo
  2. One asthma-related overnight hospitalization in the previous 12 mo
  3. One or more bursts of oral corticosteroids in the previous 12 mo
* Reside within a geographic area of the study site so that home visits are feasible.
* Have no plans to move within the upcoming 6 months
* Have insurance to cover prescription medications.
* Have a positive skin test (net wheal ≥2mm) to cat, dog, mouse, cockroach, or dust mites or have a positive cat, dog, mouse, German cockroach, or D. farinae-specific immunoglobulin E (IgE) test, as quantified using the ImmunoCAP system (≥0.35 kU/L)

Exclusion Criteria:

* Lung disease, other than asthma, that requires daily medication
* Cardiovascular disease that requires daily medication, excluding hypertension
* Taking a beta-blocker
* Allergy to dairy
* On Xolair < 5 months
* On immunotherapy and has not reached maintenance dose
* Sleeping in another home 4 or more nights/week
* Active smoker defined as a positive urine screen for high levels of urine cotinine
* Unable to access areas of home necessary to conduct extermination

Ages: 5 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 155 (Actual)
Dates: Start 2014-10-01 (Actual); Primary Completion 2018-11 (Actual); Study Completion 2018-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth C Matsui, MD MHS, Study Chair — Johns Hopkins University; Meredith McCormack, MD MHS, Principal Investigator — Johns Hopkins University; Corinne Keet, MD PHD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins University, Baltimore, Maryland, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | ECS + Medication Group | Medication Group Alone
Started | 77 | 78
Completed | 57 | 58
Not Completed | 20 | 20

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | ECS + Medication Group | Medication Group Alone | Total
Number analyzed (Participants) | 77 | 78 | 155
Age, Continuous [Mean (Standard Deviation); unit: years] | 10.1 (3.3) | 10.1 (3.3) | 10.1 (3.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31 | 30 | 61
  Male | 46 | 48 | 94
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 2 | 4
  Not Hispanic or Latino | 75 | 76 | 151
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 72 | 67 | 139
  White | 1 | 3 | 4
  More than one race | 4 | 8 | 12
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 77 | 78 | 155
The treatment step assigned [Mean (Standard Deviation); unit: score on a scale] — The controller medication treatment step that was assigned at the visit, which is based on the current controller medication treatment step and the current level of asthma control. The range is from 0-6, with 0 indicating no controller medication and 6 indicating high dose inhaled corticosteroids plus long-acting beta agonist.
  score on a scale | 4.34 (1.56) | 4.56 (1.57) | 4.45 (1.56)

OUTCOME MEASURES:

1. Primary Outcome: The Medication Treatment Step Assigned
Description: The controller medication treatment step that was assigned at the visit, which is based on the current controller medication treatment step and the current level of asthma control. The range is from 0-6, with 0 indicating no controller medication and 6 indicating high dose inhaled corticosteroids plus long-acting beta agonist.
Time Frame: 6 month clinic visit
Population: participants completing the final 6 month follow-up visit
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | ECS + Medication Group | Medication Group Alone
Number analyzed (Participants) | 63 | 62
score on a scale | 4.03 (1.91) | 4.05 (1.87)

2. Secondary Outcome: Daily Inhaled Corticosteroid Dose
Description: micrograms of inhaled corticosteroids (daily)
Time Frame: 6 months
Population: participants who completed the final follow-up visit at 6 months
Measure: Mean (Standard Deviation); unit: micrograms/day
Arm/Group | ECS + Medication Group | Medication Group Alone
Number analyzed (Participants) | 63 | 62
micrograms/day | 557.5 (347.8) | 527.7 (401.7)

3. Secondary Outcome: Exhaled Nitric Oxide
Description: Exhaled nitric oxide in parts per billion.
Time Frame: 6 months
Population: participants completing the final follow-up visit at 6 months with valid exhaled nitric oxide measurement. Not all participants had valid measures.
Measure: Median (Inter-Quartile Range); unit: parts per billion
Arm/Group | ECS + Medication Group | Medication Group Alone
Number analyzed (Participants) | 58 | 61
parts per billion | 20 [10 to 38] | 20 [8 to 52]

4. Secondary Outcome: Number of Asthma Symptom Days
Description: Number of asthma symptom days in the past two weeks will be a measure of asthma control.
Time Frame: 6 months
Population: participants who completed the final follow-up visit at 6 months.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | ECS + Medication Group | Medication Group Alone
Number analyzed (Participants) | 62 | 63
days | 2.5 (3.2) | 2.7 (3.6)

5. Secondary Outcome: Number of Asthma Exacerbations
Description: Asthma exacerbations will be assessed by number of acute visits to the emergency department (ED), hospitalizations and urgent doctor visits.
Time Frame: 6 months
Population: participants completing the 6 month follow-up visit
Measure: Number; unit: acute visits
Arm/Group | ECS + Medication Group | Medication Group Alone
Number analyzed (Participants) | 63 | 62
acute visits | 35 | 53

6. Secondary Outcome: FEV1/FVC
Description: Forced expiratory volume at one second/forced vital capacity (FEV1/FVC) will be evaluated as a continuous variable. This is a ratio without any units.
Time Frame: 6 months
Population: participants completing the 6 month follow-up visit
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | ECS + Medication Group | Medication Group Alone
Number analyzed (Participants) | 63 | 62
ratio | 79.3 (8.1) | 80.8 (8.8)

ADVERSE EVENTS:
Time Frame: During the enrollment period, approximately 7 months
Description: Hospitalizations, including asthma-related hospitalizations, were considered serious adverse events. Participants were asked at each clinic visit about adverse events.
Arm/Group | ECS + Medication Group | Medication Group Alone
All-Cause Mortality (participants affected / at risk) | 0/77 | 0/78
Serious Adverse Events (participants affected / at risk) | 2/77 | 10/78
Other Adverse Events (participants affected / at risk) | 0/77 | 0/78
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ECS + Medication Group (N=77) | Medication Group Alone (N=78)
asthma hospitalization (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 8 (11)
hospitalization (Psychiatric disorders) | 0 (0) | 1 (1)
hospitalization (Gastrointestinal disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-10-03): https://cdn.clinicaltrials.gov/large-docs/79/NCT02251379/Prot_SAP_000.pdf